CLINICAL TRIAL: NCT00099060
Title: A Phase I/II Study of GW572016 in Patients With Recurrent Malignant Glioma
Brief Title: Lapatinib in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I170; CAN-NCIC-IND170; CDR0000389155 (Other: PDQ)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2012-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult gliosarcoma; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lapatinib ditosylate — For patients receiving enzyme inducing anti-epileptic drugs (EIAEDs):
  * Phase I: starting dose for first cohort: 1000 mg GW572016 po b.i.d.; actual dose assigned at registration; intra patient dose escalation permitted ONCE in phase I patients ONLY if specified criteria met (see section 8.6).
  * Phase II: Recommended phase II dose from phase I portion of the study, given po b.i.d.
  For patients NOT receiving enzyme inducing anti-epileptic drugs (NON-EIAEDs):
  • Phase II: 750 mg GW572016 po b.i.d.
  For all patients:
  • Dose reductions as required based on adverse events.

SUMMARY:
RATIONALE: Lapatinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

PURPOSE: This phase I/II trial is studying the side effects and best dose of lapatinib and to see how well it works in treating patients with recurrent glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Phase I

* Determine the maximum tolerated dose and recommended phase II dose of lapatinib in patients with recurrent malignant glioblastoma multiforme who are taking CYP3A4 enzyme-inducing anti-epileptic drugs (EIAEDs).
* Determine the toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.

Phase II

* Determine the efficacy of this drug, in terms of objective tumor response rate, in patients who are taking EIAEDs and in those who are not taking EIAEDs.
* Correlate immunohistochemical measures of cellular proteins and receptors from tumor samples with anti-tumor activity of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is a multicenter, open-label, phase I, dose-escalation study followed by a phase II study.

* Phase I: Patients receive oral lapatinib twice daily on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of lapatinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive lapatinib as in phase I at the MTD. Patients are followed at 1 month and then periodically for survival. Patients with stable or responding disease who go off therapy are followed every 3 months for up to one year and then periodically thereafter for survival.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for the phase I portion of this study within 18 months. A total of 15-30 patients will be accrued for the phase II portion of this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioblastoma multiforme
* Recurrent or progressive disease after prior primary treatment with radiotherapy with or without adjuvant chemotherapy
* Bidimensionally measurable disease on CT scan or MRI with at least one lesion ≥ 1 cm x 1 cm
* Paraffin embedded tumor sample available
* Concurrent enzyme-inducing anti-epileptic drugs (EIAEDs) required for phase I of the study

  * Patients in phase II of the study may or may not be receiving EIAEDs

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* LVEF ≥ 50% by echocardiogram or MUGA
* No myocardial infarction within the past 6 months
* No congestive heart failure
* No unstable angina
* No active cardiomyopathy
* No cardiac arrhythmia
* No uncontrolled hypertension

Pulmonary

* No pulmonary disease requiring oxygen

Neurologic

* No preexisting peripheral neuropathy ≥ grade 3
* No history of significant neurologic disorder that would preclude study compliance or ability to give informed consent

Gastrointestinal

* No upper gastrointestinal or other conditions that would preclude compliance with oral medication
* No active peptic ulcer disease

Other

* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, curatively treated carcinoma in situ of the cervix, or other curatively treated solid tumor
* No immune deficiency
* No history of significant psychiatric disorder (e.g., uncontrolled psychotic disorders) that would preclude study compliance or ability to give informed consent
* No other serious illness or medical condition that would preclude study participation
* No known hypersensitivity to compounds of similar chemical or biological composition to lapatinib
* No active uncontrolled or serious infection
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent prophylactic filgrastim (G-CSF), sargramostim (GM-CSF), or other hematopoietic growth factors

  * Concurrent hematopoietic growth factors allowed for treatment of acute toxicity (e.g., febrile neutropenia)

Chemotherapy

* See Disease Characteristics
* No prior chemotherapy for recurrent disease
* No more than one prior chemotherapy regimen in the adjuvant setting

  * At least 6 months since prior adjuvant chemotherapy

Endocrine therapy

* Concurrent steroids allowed provided the dose is stable for at least 14 days before study entry

Radiotherapy

* See Disease Characteristics
* At least 6 weeks since prior radiotherapy

Surgery

* At least 2 weeks since prior major surgery

Other

* H2 blockers and proton pump inhibitors allowed, unless they are CYP3A4 inducers or inhibitors
* At least 7 days since prior and no concurrent administration of any of the following CYP3A4 inhibitors:

  * Clarithromycin
  * Erythromycin
  * Troleandomycin
  * Telithromycin
  * Ciprofloxacin
  * Norfloxacin
  * Itraconazole
  * Ketoconazole
  * Voriconazole
  * Fluconazole (≤150 mg/day allowed)
  * Nefazodone
  * Fluovoxamine
  * Delavirdine
  * Nelfinavir
  * Amprenavir
  * Ritonavir
  * Indinavir
  * Saquinavir
  * Lopinavir
  * Verapamil
  * Diltiazem
  * Aprepitant
  * Grapefruit or grapefruit juice
  * Bitter orange
* At least 14 days since prior and no concurrent administration of any of the following CYP3A4 inducers:

  * Rifampin
  * Rifabutin
  * Rifapentine
  * Efavirenz
  * Nevirapine
  * Hypericum perforatum (St. John's wort)
  * Modafinil
* At least 6 months since prior and no concurrent administration of amiodarone
* Antacids (e.g., mylanta, maalox, tums, rennies) must be administered ≥ 1 hour before and ≥ 1 hour after study drug
* At least 2 days since prior and no concurrent cimetidine
* No other concurrent anti-cancer agents
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-12; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Toxicity for phase I assessed by CTCAE v.3.0 MacDonald criteria | 7 years
Response for phase II | 7 years

SECONDARY OUTCOMES:
Correlative studies on archival tissue | 7 years
Pharmacokinetics | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian A. Thiessen, MD, Study Chair — British Columbia Cancer Agency
Locations (6):
- Canada (6):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec